CLINICAL TRIAL: NCT05164016
Title: Evaluating Immune Response to COVID-19 Vaccines in Patients With Cancer, Transplant or Cellular Therapy Recipients
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COVVIR
Record Dates: First submitted 2021-12-16; First posted 2021-12-20 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Hematopoietic System--Cancer; Transplant-Related Cancer; Solid Tumor Malignancy; Hematologic Malignancy; Solid Organ Transplant; Hematopoietic Cell Transplant; Cellular Therapy
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is being done because the investigators would like to learn more about how well the COVID-19 vaccine works in participants with cancer or those who have received a transplant or cellular therapy.

Primary Objective

Assess the immunogenicity to COVID-19 vaccination in patients with cancer and/or transplant and cellular therapy (TCT) recipients.

Secondary Objectives

* Evaluate the antibodies response to COVID-19 vaccination in immunocompromised patients.
* Evaluate the T cell response to COVID-19 vaccination in immunocompromised patients.

Exploratory Objectives

* Assess incidence and severity of COVID-19 infections by 6 months following immunization with a SARS CoV-2 vaccine.
* Assess the durability immune response to COVID-19 vaccination.
* Assess the immunogenicity of COVID-19 vaccination in immunocompetent children and adolescents without cancer and have not undergone transplant or received cellular therapy.

DETAILED DESCRIPTION:
The investigator will collect a blood sample (about 1 teaspoon each time) from the participant when the participant receive the COVID-19 vaccine(s) as well as an additional blood samples 6 months after the last COVID-19 vaccine.

The participant will be on the study for about 6 months after the last vaccine. After the six-month blood sample is collected, the participant will be off study.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving care at St. Jude Children's Hospital or Le Bonheur Children's Hospital
* Less than 24 years old at the time of enrollment (Day 0)
* Planning to receive a COVID-19 vaccine as part of clinical care
* Patient is one of the following:

  1. Diagnosed with a Hematological Malignancy (Group A), or
  2. Received a hematopoietic cell transplant or cellular therapy (Group B), or
  3. Diagnosed with a solid tumor malignancy (Group C).
  4. Received a solid organ transplant (Group D), or
  5. Does not have cancer and has not received any type of transplant (Group E)
* Willing and able to provide informed consent

Exclusion Criteria:

* Received a COVID-19 vaccine prior to enrollment (Day 0).

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Those who meet the Eligibility Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with immunogenicity following full vaccination (6 months after last dose). | 6 months after the last vaccine dose
  The primary endpoint is immunogenicity response following full vaccination measured at 6 months after the last vaccine dose. Immunogenicity is defined as a ≥4-fold rise in the GMT of SARS-CoV-2 binding antibody to the spike protein RBD compared to the pre-vaccine baseline level or from a non-detectable GMT at the baseline to a detectable GMT after fully vaccinated. The proportion of participants with immunogenicity following full vaccination (6 months after last dose) will be described for all enrolled patients and for each disease stratum with 95% CIs. Only patients who provide a viable blood sample to evaluate immunogenicity at these time-points following completion of vaccine series will be included in this estimation.

SECONDARY OUTCOMES:
Mean and median antibodies response to COVID-19 vaccination in immunocompromised patients at day 0, second dose, third dose, post last dose (day 180). | 6 months after the last vaccine dose
  Antibody level at each time point will be summarized with mean with standard deviation and median with range. Linear mixed effect models will be used to assess the longitudinal pattern, with appropriate data transformation if necessary.
Mean and median T cell response to COVID-19 vaccination in immunocompromised patients at day 0, second dose, third dose and post last dose (day 180). | 6 months after the last vaccine dose
  T-cell response at each time point will be summarized with mean with standard deviation and median with range. Linear mixed effect models will be used to assess the longitudinal pattern, with appropriate data transformation if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Hijano, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - Le Bonheur, Memphis, Tennessee
  - LeBonheur, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: St.Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjue.org/protocols